CLINICAL TRIAL: NCT01159132
Title: Pharmacokinetics of Low Dose Raltegravir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: National Healthcare Group Pte Ltd, Singapore (Unknown); Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HIV-NAT 127
Record Dates: First submitted 2010-06-09; First posted 2010-07-09 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: pharmacokinetics; low dose raltegravir; HIV; To study the pharmacokinetics profile of low dose raltegravir (RAL) (400mg OD and 800mg OD) and standard dose of 400mg BID in Thai HIV-infected patients.
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): RAL 400 mg OD
  Interventions: Drug: raltegravir
- 2 (Active Comparator): RAL 800 mg OD
  Interventions: Drug: raltegravir

INTERVENTIONS:
Drug: raltegravir — 12 hour PK will be done on day 1 while subjects is on stable regimen with RAL 400 mg BID. After performing intensive PK, subjects will be randomized to either group A (RAL 400 mg OD) or B (RAL 800 mg OD) for 14 days and on day 15, a second 24 hour full PK will be carried out. After the intensive PK, subjects in both the groups will switched to the other dosing regimen, group A (RAL 800 mg OD) and B (RAL 400 mg OD) for another 14 days and on day 29, the third 24 hour full PK will be carried out.

SUMMARY:
The purpose of this study is to study and compare the pharmacokinetics profile of low dose raltegravir (RAL) (400mg OD and 800mg OD) and standard dose of 400mg BID in Thai HIV-infected patients.

DETAILED DESCRIPTION:
Twenty four HIV-infected volunteers on stable doses of RAL 400 mg BID for at least 3 months and with undetectable viral load will be enrolled. On Day 1, all 24 subjects will attend the first intensive PK collection for RAL 400 mg BID and the blood samples will be drawn at T = 0.0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, and 12.0 hour post medication. All 24 subjects will be randomised (1:1) to either Group A (RAL 400 mg OD) or Group B (RAL 800 mg OD) for 14 days. On day 15, a second 24 hour intensive PK will be carried out and the blood samples will be drawn. After 2nd intensive PK, the subjects will switch to the other dosing regimen. Subjects in group A will receive RAL 800 mg OD and group B will receive RAL 400 mg OD for another 14 days. On day 29, the third 24 hour intensive PK will be carried out. After the 3rd intensive PK, all 24 subjects will be switched back to the initial regimen of RAL 400 mg BID.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Evidence of HIV infection
* Age> 18 years
* On RAL 400 mg BID containing HAART regimen with a VL < 50 copies for at least 3 months before enrollment
* Willing to adhere to the protocol requirements

Exclusion Criteria:

* Evidence of RAL resistance
* History of RAL allergy
* Use of concomitant medication that may interfere with the pharmacokinetics of RAL
* Current pregnancy or lactating or planning to get pregnant
* Active drug abuse or alcoholic
* Relevant history or current condition, illness that might interfere with drug absorption, distribution, metabolism or excretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics of RAL in Thais | 29 days
  To assess AUC, Cmax, Cmin, T 1/2, clearance of RAL at dose of 400 mg BID, 800 mg OD, 400 mg OD in Thai

CONTACTS AND LOCATIONS:
Overall Officials: Jintanat Ananworanich, MD, PhD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (1):
- HIV-NAT, Bangkok, Thailand

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org